CLINICAL TRIAL: NCT06192654
Title: Small Intestinal Submucosa Graft as an Alternative to Conventional Buccal Mucosa for Substitution Urethroplasty of Anterior Urethral Strictures
Brief Title: Small Intestinal Submucosa Graft for Repair of Anterior Urethral Strictures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xiaoyong Zeng (Other)
Responsible Party: Sponsor-Investigator, Xiaoyong Zeng, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NDXF-SIS
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Urethral Stricture, Male
Keywords: urethral stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small intestinal submucosa (SIS) graft urethroplasty (Experimental): this group will use a small intestinal submucosa graft in urethroplasty.
  Interventions: Procedure: Small intestinal submucosa (SIS) graft urethroplasty
- Autologous oral bucal mucosa graft urethroplasty (Active Comparator): this group will use an autologous oral bucal mucosa graft in urethroplasty.
  Interventions: Procedure: Autologous oral bucal mucosa graft urethroplasty

INTERVENTIONS:
Procedure: Small intestinal submucosa (SIS) graft urethroplasty — Standard technique of doing a substitution urethroplasty with no modification to the surgical steps. Instead of an autologous oral bucal mucosa graft, the small intestinal submucosa graft is sutured to the healty urethral area after incision of the urethra at the stricture location.
  Arms: Small intestinal submucosa (SIS) graft urethroplasty
Procedure: Autologous oral bucal mucosa graft urethroplasty — Standard technique of doing a substitution urethroplasty with no modification to the surgical steps. The autologous oral bucal mucosa graft is sutured to the healty urethral area after incision of the urethra at the stricture location.
  Arms: Autologous oral bucal mucosa graft urethroplasty

SUMMARY:
The field of research for this study is tissue engineering and the utilization of a small intestinal submucosa graft as a substitute biomaterial for conventional buccal mucosa in substitution urethroplasty of anterior urethral strictures.

DETAILED DESCRIPTION:
Urethral stricture refers to the abnormal narrowing of the urethral lumen resulting from fibrosis that affects the urethral epithelium and underlying corpus spongiosum. The management of urethral stricture longer than 2 cm a major therapeutic challenge in clinics. Currently available surgical techniques require harvesting of grafts from autologous sites. However, there are numerous disadvantages associated with autografts, such as limited availability and variable quality, donor site morbidity, increased risk of surgical complications; thereby the application of this method is especially limited for large defects.

The hypothesis of this study is that the small intestinal submucosa graft can be used as an alternative biomaterial to buccal mucosa for substitution urethroplasty in urethral stricture patients. The aim of this study is to assess safety and efficacy of surgical treatment of patients with anterior urethral stricture using a small intestinal submucosa graft. The follow-up time for all patients in this study was 5 years. The follow-up regimen includes retrograde and pericatheter urethrography, voiding cystourethrography, uroflowmetry, cystoscopy, and voiding symptoms monitoring. Telephone follow-up will take place in between these assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients signed informed consent form
* Patients with a single, longer than 2.0 cm and shorter than or equal to 7.0 cm anterior urethral stricture
* Patients undergoing substitution urethroplasty for urethral stricture.

Exclusion Criteria:

* Patients without surgical indication
* Subtotal and total urethral strictures
* Radiation therapy to the abdomen or pelvis
* Lichen sclerosis related strictures
* Patients with previous hypospadias repair
* Neurogenic urinary tract disorders
* Mental disorders
* Patients with a known biologic sensitivity or a cultural aversion to the use of porcine materials.
* Patients with severe dysfunction of heart, lung, liver, kidney and other important organs , endocrine system and blood system.
* Patient with malignant tumor
* Patient who cannot be regularly examined due to any circumstances
* Any clinical state which does not ensure the safe implementation of study procedure (investigator's view)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Urethral patency | 4 weeks post-surgery
  A peri-urethrogram will be performed prior to catheter removal

SECONDARY OUTCOMES:
Serious adverse events | 4 weeks post-surgery
  Frequency, type and severity of serious adverse events
Voiding symptoms | 2 months up-to 5 years post-surgery
  Participants are filling out the International Prostate Symptom Score (IPSS) questionnaire.
Urine flow | 2 months up-to 5 years post-surgery
  Participants are undergoing an uroflowmetry. This test measures the volume of urine released from the body, the speed with which it is released, and how long the release takes.
Anatomic recurrence of urethral stricture observed by cystoscopy 、 Retrograde urethrography(RUG)、 Voiding cystourethrography(VCUG) | Through study completion, an average of up to 5 years
  Full assessment of the urethral lumen after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Wuhan, Hubei, China